CLINICAL TRIAL: NCT03589001
Title: A Prospective Investigation of Osgood Schlatter With 24 Month Follow-up
Brief Title: 24 Month Follow-up of Patients With Osgood Schlatter (OSD)
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Sinead Holden, Post- Doctoral Research Fellow, Aalborg University
Other Study IDs: N-20140100-5
Record Dates: First submitted 2018-07-03; First posted 2018-07-17 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Osgood-Schlatter Disease; Apophysitis
MeSH Terms: conditions — Osteochondrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OSD: 51 adolescents with Osgood Schlatter who participated in an activity modification intervention.
  Interventions: Other: Activity modification

INTERVENTIONS:
Other: Activity modification — Activity modification, exercises and gradual return to sport

SUMMARY:
Osgood Schlatter is a common knee condition, affecting approximately 10% of adolescents. OSD is thought to be a growth related pain conditon, and thus resolve after maturation. Despite this, there a lack of prospective data investigating whether this is in fact the case.

DETAILED DESCRIPTION:
This is a prospective cohort study of 51 adolescents (aged 10-14 at baseline) with Osgood schlatter. Participants are followed for two years.

ELIGIBILITY:
Inclusion Criteria:

* 10-14 years of age
* Pain at tibial tuberosity during two or more of the following activities: Sitting with a bent knee, squatting, running, jumping or stair ambulation
* Pain during palpation of tibial tuberosity
* Knee pain for 6 weeks or more

Exclusion Criteria:

* Other knee conditions that may manifest as anterior knee pain (Patellofemoral pain, iliotibial band syndrome, sinding-larson-johanson disease).
* Previous surgery
* Pain from the hip or back that interferes with activities of daily living.
* Habitual patella luxations
* Clinical suspicion of meniscal lesion

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescents aged 10-14 years old diagnosed with Osgood Schlatter
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Current knee pain | 24 months
  Participants self-report if they still have knee pain

SECONDARY OUTCOMES:
Pain intensity | 24 months
  Worst pain in the previous week measured on a visual analogue scale (VAS) from 'no pain' to 'worst imaginable pain'
Pain frequency | 24 months
  Frequency of knee pain divided into (almost daily, several times per week, weekly, monthly, rarely, never)
Duration of being pain-free | 24 months
  Those who no longer have knee pain will be asked how long since their knee pain resoved
Medical attention | 24 months
  Participants will be asked to report if they sought medical attention outside of the intervention
Use of pain killers | 24months
  Participants will be asked if they use painkillers to manage their knee pain (y/n). If yes, they will be asked how often.
knee injury and osteoarthritis outcomes score (KOOS) sport and activity subscale | 24 months
  knee injury and osteoarthritis outcomes score (KOOS) subscale sport and activity. Minimum 0 points, maximum 100points, with 100 points being the best possible score.
Sports participation | 24 months
  Participants will report if they participate in sport. If yes how often and how much/week. They will also report if they have reduced sports participation due to knee pain.
Health Related quality of life | 24 months
  Health related quality of life assessed by EQ 5D 3L Y (EuroQol, 5 dimensions, 3 levels for youth). Minimum 0, maximum 1, with higher values indicating higher quality of life.
Sleep | 24 months
  Participants will be asked if they find it hard to sleep because of their knee pain (not at all, some nights, most nights).

CONTACTS AND LOCATIONS:
Locations (1):
- Research Unit for General Practice in Aalborg, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon reasonable request, inline with Data Protection procedures